CLINICAL TRIAL: NCT00036985
Title: A Randomized Pivotal Clinical Trial To Assess The Efficacy Of Pre-operative Focused Microwave Thermotherapy Treatment Combined With Pre-operative Chemotherapy For Cytoreduction Of Advanced Breast Cacer In Intact Breast
Brief Title: Combination Chemotherapy With or Without Microwave Thermotherapy Before Surgery in Treating Women With Locally Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Imunon (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069346; CELSION-10200201; OU-09533
Record Dates: First submitted 2002-05-13; First posted 2003-01-27 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2004-07

CONDITIONS: Breast Cancer
Keywords: stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Doxorubicin; Neoadjuvant Therapy

INTERVENTIONS:
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Procedure: thermal ablation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Microwave thermotherapy kills tumor cells by heating them to several degrees above body temperature. Combining chemotherapy with microwave thermotherapy before surgery may shrink the tumor so that it can be removed during surgery.

PURPOSE: Randomized phase II trial to compare the effectiveness of combination chemotherapy with or without microwave thermotherapy before surgery in treating women who have locally advanced breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the safety and efficacy of neoadjuvant therapy comprising cytoreductive doxorubicin and cyclophosphamide with or without focused microwave thermotherapy in women with locally advanced breast cancer in an intact breast.
* Evaluate percentage of patients who achieve at least 85% pathological cell death after treatment with focused microwave thermotherapy.
* Compare clear pathology tumor margins and reduction of second incision rates in patients treated with these regimens.
* Compare the amount of surgically removed breast and tumor tissue in patients treated with these regimens.
* Compare the measurement of the extent of tumor margins in patients treated with these regimens.
* Compare the reduction of tumor size in patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to tumor size (T2 vs T3). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive cyclophosphamide IV over 15 minutes and doxorubicin IV over 15 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of unacceptable toxicity.

During courses 1 and 2 only, patients undergo focused microwave thermotherapy on day 1 of chemotherapy (or within 36 hours after chemotherapy). Patients undergo ultrasound-guided placement of a microwave sensor and a temperature probe (before or after compression of the breast) and external placement of 2 large opposing microwave emitters and up to 7 skin temperature sensors on the compressed breast. Patients then receive focused microwave thermotherapy that slowly heats the primary breast tumor and deep proximal breast tissue. In the absence of any unacceptable toxicity, a target tumor temperature of 43-47° C is reached and maintained for an equivalent thermal dose of 80-120 minutes.

* Arm II: Patients receive chemotherapy only as in arm I. Within 60 days after completion of thermochemotherapy or chemotherapy alone, patients in both arms undergo total mastectomy, partial mastectomy, or other breast-conserving surgery, as appropriate. At the discretion of the physician, beginning after completion of chemotherapy, patients in both arms who are estrogen receptor positive may receive oral tamoxifen. Within 4 weeks after completion of chemotherapy and surgery, eligible patients in both arms also undergo radiotherapy to the breast and lymph nodes.

Patients are followed at 30 and 90 days.

PROJECTED ACCRUAL: A total of 280-312 patients (140-156 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed locally advanced primary breast cancer

  * Stage III (T2-3, N2-3) disease
  * Diagnosis not made by lumpectomy or incisional biopsy
* Currently a candidate for mastectomy and neoadjuvant chemotherapy
* Primary tumor measurable by breast ultrasound and clinical exam
* No bilateral breast cancer
* No high probability for extensive intraductal in situ disease
* No clinical fixation to the pectoralis major muscle or skin
* No involvement of the nipple
* No inflammatory breast cancer
* No multicentric disease
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Karnofsky 70-100%

Life expectancy:

* At least 6 months

Hematopoietic:

* Platelet count at least 100,000/mm^3 (no thrombocytopenia)
* No bleeding disorders

Hepatic:

* PT and PTT less than 1.5 times normal
* INR less than 1.5 times normal
* Bilirubin no greater than 2.0 mg/dL
* Transaminases no greater than 2 times normal
* No coagulopathy
* No liver disease

Renal:

* BUN less than 30 mg/dL OR
* Creatinine less than 1.9 mg/dL
* No renal insufficiency

Cardiovascular:

* No clinically significant heart disease
* No pacemakers or defibrillators

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 effective methods of contraception
* No breast implants
* No prior collagen vascular disease
* No concurrent mental condition that would preclude study
* No contraindications to chemotherapy
* Able to tolerate prone position and breast compression

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Other:

* No prior participation in this study
* More than 30 days since participation in another clinical trial
* No concurrent participation in another clinical trial
* No concurrent anticoagulants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-08

CONTACTS AND LOCATIONS:
Overall Officials: William E. Gannon, MD, Study Chair — Imunon
Locations (7):
- United States (7):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - St. Joseph Hospital Regional Cancer Center - Orange, Orange, California
  - Comprehensive Breast Center of Coral Springs, Coral Springs, Florida
  - Oklahoma University Medical Center at University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mroz-Baier Breast Care Center, Memphis, Tennessee
  - Breast Care Specialists, P.C., Norfolk, Virginia
  - Tacoma, Washington